CLINICAL TRIAL: NCT00506454
Title: A Phase II, Double-Blind, Placebo-Controlled, Randomized Study of the Effects of a Lipid Emulsion (Lipidose) on Endotoxin Levels in Patients on Chronic Hemodialysis
Brief Title: Lipid Infusion in Dialysis Patients With Endotoxemia
Acronym: LIPIDOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sepsicure (Industry)
Collaborators: The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S201
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Fatigue; End Stage Renal Disease (ESRD)
Keywords: Fatigue; Hemodialysis; Endotoxemia; Phospholipid; Emulsion
MeSH Terms: conditions — Fatigue; Kidney Failure, Chronic; Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipidose (Active Comparator): Dosage of 1.5 mL/kg of Lipidose over a 2-hour period.
  Interventions: Drug: Lipidose
- Placebo (Placebo Comparator): Dosage of 1.5 mL/kg of Placebo over a 2-hour period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lipidose — Over the course of 2 weeks, immediately following subject's three (Monday/Wednesday/Friday (M/W/F)) normal dialysis treatments, based on subject's current weight, subject will receive 1.5 mL/kg of Lipidose over a 2-hour period.
  Other Names: GR270773
  Arms: Lipidose
Drug: Placebo — Over the course of 2 weeks, immediately following subject's three (M/W/F) normal dialysis treatments, based on subject's current weight, subject will receive 1.5 mL/kg of placebo over a 2-hour period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a phospholipid emulsion is effective in the treatment of chronic endotoxemia in hemodialysis patients.

DETAILED DESCRIPTION:
Over 70% of dialysis patients suffer chronically from severe fatigue and tiredness. A possible inciting factor may be high levels of circulating endotoxin, which is well-established as a potent stimulator of inflammatory cytokine release.

The source of increased endotoxin in dialysis patients remains unclear, with the most popular hypotheses including back-diffusion of bacterial products from nonsterile dialysate and translocation of bacterial products across what in most dialysis patients is an edematous gut wall. This endotoxin does not appear to be associated with the dialysis procedure itself and indeed, appears to be cleared with some efficiency by the procedure. However, by the next dialysis treatment, endotoxin levels rise rapidly to levels that are in some cases significantly higher than even those measured (via EAA) in patients suffering from septic shock. Although the mechanisms by which dialysis patients tolerate these high endotoxin levels without hemodynamic collapse are not understood, high levels have been shown by The Rogosin Institute to significantly correlate with patient fatigue.

Given the potent ability of endotoxin to induce expression of inflammatory cytokines (which in turn are likely responsible for the debilitating symptoms of fatigue and malaise that afflict the majority of the dialysis population), it is logical that binding and inactivation of endotoxin may lead to improved clinical outcomes. Unfortunately, there are no products currently approved for this purpose in dialysis patients.

One approach to this problem may be to augment the endogenous systems for endotoxin inactivation. For example, it has been suggested that the various serum lipoprotein fractions may in fact be a physiologic "sink" for endotoxin (and other toxins) via binding with surface phospholipids. Therefore, dialysis patients, who as a population are characterized with hypocholesterolemia and hypolipoproteinemia, are particularly at risk for the deleterious effects of endotoxemia.

This has led to the development of "LIPIDOSE," a protein-free phospholipid emulsion. The proposed mechanism of action of this compound is via remodeling of the infused phospholipids into lipoproteins, thereby increasing lipoprotein and phospholipid content and facilitating greater endotoxin binding and neutralization. "LIPIDOSE" has undergone extensive testing in both animals and humans, and has been found to significantly increase serum phospholipid and lipoprotein concentrations, improve survival in a lethal animal model of septic peritonitis, and mitigate the symptoms of endotoxemia in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. On hemodialysis for ≥ 3 months.
2. Provided written and dated informed consent.
3. Meets the following lab parameters on Screening labs:

   * Serum albumin > 2.5 g/dL;
   * Serum total cholesterol > 95 mg/dL;
   * Serum High-Density Lipoprotein (HDL) > 20 mg/dL;
   * Serum hemoglobin ≥ 11 g/dL;
   * Serum transaminases < 2x the upper limit of normal.
4. Has had a dialysis adequacy level (KT/V) greater than 1.3 for 2 months prior to screening.
5. Has a vitality score of ≤ 16 at time of screening.

Exclusion Criteria:

1. Currently participating in or has participated in an investigational drug or medical device study within 30 days or five half-lives, whichever is longer, prior to enrollment in this study.
2. Pregnant, breast-feeding or female of childbearing potential who does not agree to remain abstinent or to use an acceptable contraceptive regimen (oral contraceptive, double-barrier method, or abstention from sexual relations) during the study period.
3. Has any of the following laboratory abnormalities when screened:

   * Serum haptoglobin below the lower limit of normal;
   * Lactate dehydrogenase (LDH) > 300 U/L;
   * Low-Density Lipoprotein (LDL) > 190 mg/dL;
   * Fasting (8 hours, water only) triglyceride level > 300 mg/dL;
   * Serum phospholipid level > 500 mg/dL.
4. Has an EAA level < 0.6 Endotoxin Activity (EA) at screening.
5. Has prolonged heart wave (QT) interval (as defined by corrected QT (QTc) > 460 msec in males and > 470 msec in females) on screening electrocardiogram (ECG).
6. Has a history of allergic reaction to eggs (or egg products), soybeans, Intralipid, or any component of "LIPIDOSE".
7. Has had a recent hospitalization (within the last 30 days) or has other acute illness.
8. Deemed not medically or psychiatrically stable for the study (in opinion of investigator or the subject's primary nephrologist).
9. Currently on any of the following medications: (a) medications known to cause QT prolongation; (b) parenteral nutrition supplements (e.g., Intralipid); (c)amphotericin; (d) liposomal amphotericin; (e) amphotericin B lipid complex; or (f) coumadin.
10. Has known preexisting systolic dysfunction (as defined by previous echocardiogram with ejection fraction (EF) < 35%).
11. Currently receiving one of the following prohibited concomitant medications; parenteral nutrition supplements containing lipid "emulsion" (e.g., Intralipid), amphotericin, liposomal amphotericin, or amphotericin B lipid complex.
12. Has a known active hemolytic disease; immune hemolytic anemias, hemoglobinopathies (sickle cell anemia and thalassemia major) or is known or believed to suffer from hereditary spherocytosis or S.E. Asian elliptocytosis.
13. Has a known bone marrow disorder of inadequate red cell production (e.g., aplastic anemia, myelodysplasia).
14. Has known current alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Bologa, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- Rogosin Manhattan Dialysis Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Participants receiving the active drug.
- Placebo: Participants receiving the placebo.
Period: Overall Study
Arm/Group | Active | Placebo
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 49.3 (11.57) | 55.5 (7.88) | 52.4 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Endotoxin Levels.
Description: The number of participants whose post-hemodialysis endotoxin (as measured by Endotoxin Activity Assay (EAA)) was less than their pre-hemodialysis endotoxin.
Time Frame: Baseline and at 4 weeks
Measure: Number; unit: Participants
Groups:
- Treatment: Participants receiving the active drug.
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
There was no significant difference between endotoxin activity assay values in the active versus placebo recipients in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No